CLINICAL TRIAL: NCT04280822
Title: A Phase III, Randomized Controlled Study of Neo-adjuvant Toripalimab (JS001) in Combination With Chemotherapy Versus Neo-adjuvant Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neo-adjuvant Immunochemotheray Versus Neo-adjuvant Chemotherapy for Resectable Esophageal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCHTOG1909
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Cancer; Surgery; Neoadjuvant Treatment; Survival
Keywords: Neoadjuvant chemotherapy; Neoadjuvant immunochemotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant immunochemotherapy (Experimental): Neo-adjuvant chemotherapy(cisplatin and paclitaxel):
  Paclitaxel, 175mg/m2, d1, Cisplatin, 75mg/m2, d1, 3 week, 2 cycles. JS001, 240mg ivgtt, d3, >30min, 3week, 2 cycles
  Surgery:
  2-3weeks after Neo-adjuvant chemotherapy Surgeons: the operation shall be performed by senior thoracic surgeons. Try to achieve the consistency of operation quality.
  Operation: the thoracic esophagectomy must be through right thoracic cavity. (open and minimally invasive McKeown or Ivor Lewis). Total two-field lymphadenectomy (right and left recurrent laryngeal nerve lymph nodes must be included).
  After surgery/ maintain period:
  JS001, 240mg ivgtt, d3, >30min, 3week (8 cycles at most)
  Interventions: Drug: Neoadjuvant immunochemotherapy
- Neoadjuvant chemotherapy (Active Comparator): Neo-adjuvant chemotherapy(cisplatin and paclitaxel):
  Paclitaxel, 175mg/m2, d1, Cisplatin, 75mg/m2, d1, 3 week, 2 cycles.
  Surgery:
  2-3weeks after Neo-adjuvant chemotherapy Surgeons: the operation shall be performed by senior thoracic surgeons. Try to achieve the consistency of operation quality.
  Operation: the thoracic esophagectomy must be through right thoracic cavity. (open and minimally invasive McKeown or Ivor Lewis). Total two-field lymphadenectomy (right and left recurrent laryngeal nerve lymph nodes must be included).
  Interventions: Drug: Neoadjuvant immunochemotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — Neo-adjuvant chemotherapy(cisplatin and paclitaxel):
  Paclitaxel, 175mg/m2, d1, Cisplatin, 75mg/m2, d1, 3 week, 2 cycles. JS001, 240mg ivgtt, d3, >30min, 3week, 2 cycles
  Surgery:
  2-3weeks after Neo-adjuvant chemotherapy Surgeons: the operation shall be performed by senior thoracic surgeons. Try to achieve the consistency of operation quality.
  Operation: the thoracic esophagectomy must be through right thoracic cavity. (open and minimally invasive McKeown or Ivor Lewis). Total two-field lymphadenectomy (right and left recurrent laryngeal nerve lymph nodes must be included).
  After surgery/ maintain period:
  JS001, 240mg ivgtt, d3, >30min, 3week (8 cycles at most)

SUMMARY:
The effect of neo-adjuvant immunochemotherapy on survival of patients with thoracic esophageal squamous cell carcinomas remains unknown. One of our objectives is to evaluate whether the neo-adjuvant immunochemotherapy Toripalimab (JS001) with cisplatin and paclitaxel followed by right thoracic approach esophagectomy with total 2-field lymph node dissection improves the overall survival of thoracic esophageal cancer patients versus neo-adjuvant chemotherapy.

DETAILED DESCRIPTION:
The effect of immunochemotherapy in second line treatment of esophageal cancer got a positive results in the world. We tried to apply the immunotheray in resectable esophageal cancer and have planed this phase III clinical trials. The optimal management of resectable esophageal squamous cell carcinomas may have a new chapter in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of local advance squamous cell thoracic esophageal carcinoma of Stage (T1N1-3 or T2-3N0-3 M0), (8th Union for International Cancer Control, UICC-TNM).
2. No metastatic lymph node in cervical by color doppler sonography.
3. Patients must not have received any prior anticancer therapy of esophageal carcinoma.
4. Age ranges from 18 to 75 years.
5. Without operative contraindication.
6. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney, total bilirubin（TBIL）≤1.5N, aspartate aminotransferase (AST)≤2.5N, alanine aminotransferase(ALT)≤2.5N, prothrombin time(PT)≤1.5N, and activated partial thromboplastin time(APTT) is in normal range, endogenous creatinine clearance rate(CRE)≤1.5N.
7. Patients must not have diagnosed with other cancer and must not received any prior anticancer therapy except prostatic cancer with more than 5 years disease-free survival(DFS).
8. expected R0 resection.
9. ECOG 0～1.
10. Patients should agree to use contraceptive measures during the study period and within 6 months of the end of the study. Women must be non-lactation.
11. Signed informed consent document on file. 10. .

Exclusion Criteria:

* 1. Multiple primary cancer. 2.Patients with infections disease that require treatment 3.Patients who need continuous hormone treatment 4.unstable angina within 3 months, myocardial infarction within 6 months 5.psychopath 6.Patients with concomitant hemorrhagic disease. 7.Any unexpected reason for patients can't get operation 8.Inability to use gastric conduit after esophagectomy because of a prior surgery.

  9.Pregnant or breast feeding 10.Patients are diagnosed or suspected to be allergic to cisplatin or Paclitaxel.

  11.Bronchial asthma who requires intermittent use of bronchodilators or medical interventions 12.Due to co-existing diseases, the immunosuppressant was used. And the dosage of immunosuppressant was more than 10mg/ day orally and more than 2 weeks before enrollment 13.Abnormal coagulation function (PT>16s, APTT>53s, TT>21s, Fib<1.5g/L), tendency of bleeding or receiving thrombolysis or anticoagulant therapy 14.Previous or present pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, lung function severely impaired 15.Autoimmune diseases, immune deficiency, organ transplantation； 16.Hepatitis b/c patients。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | The date from the beginning of randomization to the date of first record. 3 years EFS
  The date from the beginning of randomization to the date of first record of unresectable disease, distant metastases, local recurrences of any causes, and death of any cause.
Event-free survival (EFS) | The date from the beginning of randomization to the date of first record. 5 years EFS
  The date from the beginning of randomization to the date of first record of unresectable disease, distant metastases, local recurrences of any causes, and death of any cause.

SECONDARY OUTCOMES:
pCR | within 14 working days after operation
  pathological complete response rate
DFS | 3 years DFS
  Disease free survival
DFS | 5 years DFS
  Disease free survival
OS | 3 years OS
  Overall survival rate
OS | 5 years OS
  Overall survival rate
ORR | 3-4 weeks after the last cycle of neoadjuvant treatment
  The Overall Response Rate. ORR=CR+PR. Criteria: Response Evaluation Criteria in Solid Tumors, RECIST.
R0 resection rate | within 14 working days after operation
  the complete resection rate of all tumor under microscope
MPR | within 14 working days after operation
  MPR rate was defined as the percentage of patients who achieved a major pathological response (residual tumor ≤10%)
EORTC QLQ-C30 | before surgery, 1month, 3 months, 6 months, 9 months, 1 year after operation
  EORTC QLQ-C30 repeated measurement model
EORTC QLQ-OES18 | before surgery, 1month, 3 months, 6 months, 9 months, 1 year after operation
  EORTC QLQ-OES18 repeated measurement model
NRS-2002 | before surgery, 1month, 3 months, 6 months, 9 months, 1 year after operation
  NRS-2002 repeated measurement model

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, PhD, MD, Principal Investigator — Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university
Locations (1):
- Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Zheng Y, Liu XB, Sun HB, Xu J, Shen S, Ba YF, Yan M, Qin Z, Liu BX, Wang ZF, Liu SL, Zhang RX, Chen PN, Liang GH, Yuan D, Li ZX, Liu Q, Wang HR, Li HM, Lv H, Ma X, Zhu J, Yu YK, Xing WQ; written on Henan Cancer Hospital Thoracic Oncology Group (HCHTOG). A phase III study on neoadjuvant chemotherapy versus neoadjuvant toripalimab plus chemotherapy for locally advanced esophageal squamous cell carcinoma: Henan Cancer Hospital Thoracic Oncology Group 1909 (HCHTOG1909). Ann Transl Med. 2021 Jan;9(1):73. doi: 10.21037/atm-20-5404. PMID 33553366